CLINICAL TRIAL: NCT04750187
Title: Effects of Hypo-pressive Abdominal Exercise on Inspiratory Muscle Strength, Diaphragm Thickness and Pain in Patients With Chronic Nonspecific Low Back Pain
Brief Title: Hypo-pressive Abdominal Exercise on Inspiratory Muscle Strength, Diaphragm Thickness and Pain in Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFV_1/2021
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypo-pressive abdominal exercise program (Experimental)
  Interventions: Other: Hypo-pressive abdominal exercise intervention
- No training program (No Intervention)

INTERVENTIONS:
Other: Hypo-pressive abdominal exercise intervention — An 8-week hypo-pressive abdominal exercise program
  Arms: Hypo-pressive abdominal exercise program

SUMMARY:
The purpose of this study will be to assess the effects of an 8-week hypo-pressive abdominal exercise program on Inspiratory muscle strength, diaphragm thickness, pressure pain threshold and disability in patients with non-specific chronic low back pain. A randomized clinical trial will be carried out. A total sample of 40 patients with non-specific chronic low back pain will be recruited and divided into 2 groups including an experimental group (n=20) which will receive an 8-week hypo-pressive abdominal exercise program and a control group (n=20) which will not receive any training program. Inspiratory muscle strength, diaphragm thickness, pressure pain threshold and disability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-specific low back pain

Exclusion Criteria:

* Congenital diseases
* Rheumatic or neuro-muscular diseases
* Respiratory conditions
* Surgery
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | Change from baseline inspiratory muscle strength at 8 weeks
  Inspiratory muscle strength will be measured in % by a POWER-breathe device

SECONDARY OUTCOMES:
Diaphragm muscle thickness | Change from baseline diaphragm muscle thickness at 8 weeks
  Diaphragm muscle thickness will be measured in mm by an ultrasound device
Pressure pain threshold | Change from baseline pressure pain threshold at 8 weeks
  Pressure pain threshold will be measured in kg/cm2 by an algometer
Disability | Change from baseline disability at 8 weeks
  Pain-related disability score will be measured by the Roland-Morris Disability Questionnaire. Total score ranges from 0 to 24. Higher scores represent higher levels of pain-related disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calvo-Lobo C, Almazan-Polo J, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P, Rodriguez-Sanz D, Lopez-Lopez D. Ultrasonography comparison of diaphragm thickness and excursion between athletes with and without lumbopelvic pain. Phys Ther Sport. 2019 May;37:128-137. doi: 10.1016/j.ptsp.2019.03.015. Epub 2019 Mar 28. PMID 30954705